CLINICAL TRIAL: NCT04551651
Title: AppReminders Trial - A Pilot Feasibility Trial of a Memory Aid App for People With Acquired Brain Injury
Brief Title: AppReminders - A Pilot Feasibility Trial of a Memory Aid App for People With Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN19NE236
Record Dates: First submitted 2019-05-24; First posted 2020-09-16 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Acquired Brain Injury
Keywords: Assistive Technology for Cognition; Neuropsychological Rehabilitation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ApplTree reminder app intervention (Active Comparator): A reminding app developed with features that, based on previous research, will increase use and ease of use for individuals with ABI when setting smartphone reminders.
  Interventions: Device: ApplTree
- Google Calendar reminder app intervention (Active Comparator): A widely available calendar app that can be used to set reminders.
  Interventions: Device: Google Calendar

INTERVENTIONS:
Device: ApplTree — App downloaded on the participants phone, a short video tutorial session to explain use, and technical support throughout trial period.
  Arms: ApplTree reminder app intervention
Device: Google Calendar — App downloaded on the participants phone, a short video tutorial session to explain use, and technical support throughout trial period.
  Arms: Google Calendar reminder app intervention

SUMMARY:
People with brain injury commonly experience difficulties with memory, concentration, attention and judgement, meaning that important everyday actions and tasks are not carried out or not completed, limiting the ability to live independently. Technology-based solutions, including smartphone applications, can help by providing prompts about intended actions at the correct time. However, memory and attention impairments mean people forget to set reminders or fail to set them accurately (e.g. setting the wrong time/date for events). Using co-design methods with prospective users, the investigators developed ApplTree, a smartphone reminding application with design features that can be personalised to individuals. ApplTree prompts reminder setting, supports reminder entry to improve accuracy, and delivers users with prompts at the appropriate times. A pilot randomised controlled trial will be conducted to provide crucial information to inform a future larger scale efficacy trial of ApplTree as an intervention to support memory in people with acquired brain injury.

DETAILED DESCRIPTION:
Rationale Brain injury is a leading cause of disability in Scotland. The British Society of Rehabilitation Medicine reports the prevalence of head injury in the UK to be 300 per 100,000 and the prevalence of disabled survivors of brain injury is 100-150 per 100,000. A particularly high prevalence of disability following hospitalisation for brain injury has been reported in Scotland (4.5 times higher than the Department of Health prevalence estimate).

People with brain injury commonly experience difficulties with memory, concentration, attention and judgement, meaning that important everyday actions and tasks are not carried out or not completed, limiting the ability to live independently. Technology-based solutions, including smartphone applications, can help by providing prompts about intended actions at the correct time. However, memory and attention impairments mean people forget to set reminders or fail to set them accurately (e.g. setting the wrong time/date for events). Using co-design methods with prospective users, the investigators developed ApplTree, a smartphone reminding application with design features that can be personalised to individuals. ApplTree prompts reminder setting, supports reminder entry to improve accuracy, and delivers users with prompts at the appropriate times. The investigators wish to find out if such an intervention can improve the everyday memory performance of individuals with memory difficulties following acquired brain injury compared to an off-the-shelf reminding app (Google Calendar). During this project a pilot randomised controlled trial will be conducted to provide crucial information to inform a future larger scale efficacy trial of ApplTree as an intervention to support memory in people with acquired brain injury.

ApplTree app The investigators designed ApplTree with features that our research suggests can help support independent use and increase the efficacy of prompting technology interventions, and which can be personalised according to need and preference.

User Interface (UI) Type: ApplTree has the option of a traditional 'broad-shallow' UI or a 'narrow-deep' UK. The 'narrow-deep' UI has several screens but little information on each screen. Previous research has indicated that this is preferable for people with cognitive impairments when searching for content online compared to the alternative, and more common, 'broad-shallow' UI that contains lots of information on each screen but a small number of screens.

Unsolicited Prompts (UPs): ApplTree provides periodic prompts to encourage the user to set reminders. This is helpful if people have self-monitoring, initiation or mood problems that are common after neurological injury. The investigators investigated UP's previously using a single case experimental design (n=3). Participants set more reminders when receiving UPs illustrating their potential to increase reminder setting. More investigation is needed to understand how they influence acceptability.

Carer Support in App: Reminding software that allows input from carers can be effective as a memory aid. ApplTree allows carer input so that carers can, when appropriate, set reminders and send prompts to the patient.

Scientific justification Technologies that send timely prompts to people about everyday activities are an effective, low cost solution to support people with cognitive impairments after brain injury. Our systematic review and meta-analysis found that prompting technology improves memory performance for people with memory difficulties vs. practice as usual or a paper diary/calendar (d = 1.27, large effect size, n=147). Reminding technology can also reduce the burden on caregivers. This potential positive impact will only be seen in practice if people have access to this technology (e.g. as part of their clinical rehabilitation). The positive impact of reminding technology use will be greater if people are able to use the technology independently when it is provided, and if the technology meets the individual needs of the users. Our systematic review found few papers that investigated smartphone apps (the state-of-the-art technology for delivering prompts) delivered through a clinical service. Furthermore, only three studies asked participants to set reminders independently, which is crucial to increasing functional independence. Our research with smartphone users with ABI has highlighted that memory and attention difficulties prevent people from making effective use of reminding apps. Due to cognitive impairments impacting usability, those who could benefit most from reminding technology are the people for whom it is least accessible. This may explain why uptake of reminding technology is currently low. There is, however, insufficient evidence regarding the best user interface design for apps to ensure that people with cognitive impairments are able to use them independently. It is also unknown whether it is feasible and effective to introduce an app with these features to patients through clinical services. Answering these questions is vital for this intervention to improve independent functioning and alleviate caregiver burden.

This project will build on extensive previous work developing ApplTree - smartphone reminding software with personalisable features, specifically designed for people with brain injury to improve everyday functioning. Interventions that can be tailored to individuals' needs are consistent with the drive towards personalised/ stratified medicine and treatment delivery. The investigators will undertake a user study and a pilot randomised controlled trial that will underpin a large-scale RCT to examine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Acquired brain injury
* Self or other reported memory difficulties resulting from an acquired brain injury

Exclusion Criteria:

* Inability to provide informed consent for research participation
* Does not own a smartphone compatible with ApplTree and Google Calendar
* Inadequate writing or reading (English) which would impair comprehension and performance of experimental tasks, and / or answering of questionnaires.
* Inability to verbally communicate adequately in an experimental setting
* Severe physical or sensory disability which would prevent any attempt at using a typical smartphone device (e.g. paralysis of both upper limbs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment | 9 months
  The number of service users who take part in the trial
Attrition to trial sessions | 12 months
  Proportion of those randomised that attended the first, second and third follow-up sessions
Adherence to intervention | 12 months
  Proportion of people using Google Calendar or ApplTree at least once during each of the three follow-up weeks during the intervention phase (weeks 10, 11 and 12)

SECONDARY OUTCOMES:
Memory performance | 12 months
  Mean and standard variation of the difference between individual's memory performance in baseline phase (no intervention) and intervention phases (either ApplTree or Google Calendar)
Experiences of using memory apps | 12 months
  Feedback from participant's about their experiences in the trial and using the apps
Factor that may influence intervention delivery - technical help | 12 months
  a) number of times each participant asked for technical help, b) who was asked to solve each issue, c) who was able to solve this technical issue d) a short description of what the problem was
Factor that may influence intervention delivery - time required for support | 12 months
  The amount of the clinician's and researcher's time spent helping with technical issues outside of the main study sessions
Factor that may influence intervention delivery - learnability of app interventions | 12 months
  the number of times each participant had to do the assessment questions before they received a high enough score to end the intervention session. Pass mark is 60% of the information correctly entered.
Factor that may influence intervention delivery - neuropsychological profile | 12 months
  • All participants will be given four cognitive scores based on the measures provided; a memory, executive function, attention and combined 'overall cognition' score (the mean of memory, attention and executive function measures). Scaled scores or percentile rank scores will be used. Higher scores on these tests mean better cognitive ability.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Evans, Principal Investigator — University of Glasgow
Locations (4):
- United Kingdom (4):
  - Acquired Brain Injury (ABI) service, West Dun HSPC Cairnmhor Resource Centre, Joint Hospital Campus, Glasgow, Dunbartonshire
  - Community treatment Centre for Brain Injury, West Glasgow ACH Dalnair Street, Glasgow, Glasgow City
  - Quarriers Renfrewshire Acquired Brain Injury service, Paisley, Renfrewshire
  - Graham Anderson House, Springburn Road, Springburn, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided